CLINICAL TRIAL: NCT02276677
Title: Oxytocin Effects on Food Motivation Pathways
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Austen Lawson, Assistant Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SPID 1127
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): Oxytocin 24 IU x 1
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo 24 IU x 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Single dose, intranasal
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — Single dose, intranasal
  Arms: Placebo

SUMMARY:
Oxytocin is a peptide hormone produced in the brain that regulates food intake. However, the mechanisms for this effect in humans is not yet clear.

In this study, the investigators will therefore examine the effect of a single dose of intranasal oxytocin (compared to placebo) on levels of appetite-regulating hormones and functional magnetic resonance imaging activation of areas of the brain involved in food motivation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old
* BMI 25-40
* Regular breakfast eater (at least 4 times per week)
* Stable weight within the past three months

Exclusion Criteria:

* Psychiatric disease, use of psychotropic medications
* History of eating disorder
* History of excessive exercise within the last three months (having run more that 25 miles in any one week or having exercised more than ten hours in any one week)
* History of diabetes mellitus
* Active substance abuse
* Hematocrit lower than the normal range
* Gastrointestinal tract surgery (including gastrectomy, gastric bypass surgery, and small or large bowel resection)
* History of cardiovascular disease (such as hypertrophic cardiomyopathy, valvular heart disease, coronary heart disease, or coronary artery spasms)
* Untreated thyroid disease
* Tobacco use
* Cardiac pacemaker, surgical aneurysm clips, neurostimulator, implanted pumps, metal fragments in body/eyes, nitroglycerin patch, severe claustrophobia

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in functional magnetic resonance imaging activation of food motivation brain regions | Functional magnetic resonance imaging at T60 min after oxytocin/placebo

SECONDARY OUTCOMES:
Change in hormone levels (cholecystokinin, glucagon-like peptide-1) | Blood draws at T0, T30, T60, T120 min after oxytocin/placebo

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided